CLINICAL TRIAL: NCT01053429
Title: Post-Marketing Surveillance (PMS) Study to Evaluate Safety and Efficacy of Zeldox Capsule
Brief Title: A Non-Interventional Post-Marketing Surveillance Study to Evaluate the Safety and Efficacy of Zeldox Capsule
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281140
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Regulatory Post-Marketing Surveillance; Regulatory Pharmacovigilance; ziprasidone
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational cohort
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — This is a non-interventional, pharmacovigilance study, therefore patients are on ziprasidone as prescribed by their doctor.
  Other Names: Geodon, Zeldox

SUMMARY:
This is a regulatory-required non-interventional pharmacovigilance study exploring the safety profile of ziprasidone HCL monohydrate 20mg, 40mg, 60mg, 80mg in the real world patient population, thus, safety (and/or efficacy) signals will be checked at every visit during the contracted study period until the maximum study end date, per the protocol, of April 2010.

DETAILED DESCRIPTION:
All patients diagnosed with schizophrenia or acute manic or mixed episodes associated with bipolar disorder, with or without psychotic features will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia

Exclusion Criteria:

* Patients who have known hypersensitivity to any ingredient of the product
* Patients who have had a recent acute myocardial infarction
* Patients who have uncompensated heart failure
* Patients who have conditions with a potential to increase QT interval (QT-interval prolongation or history of QT prolongation; congenital long QT syndrome; use with other drugs known to increase the QT interval; arrhythmias treated with class I and III antiarrhythmic drugs)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with schizophrenia or acute manic or mixed episodes associated with bipolar disorder, with or without psychotic features will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3391 (Actual)
Dates: Start 2005-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281140&StudyName=A%20Non-Interventional%20Post-Marketing%20Surveillance%20Study%20to%20Evaluate%20the%20Safety%20and%20Efficacy%20of%20Zeldox%20Capsule

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric patients <18 years of age (N=105) were enrolled in error by some sites and were subsequently reported as protocol violations. Given that the objective of this Non-interventional study was to observe the safety and efficacy of Zeldox in real life, the data collected from these participants was included in the safety and efficacy analyses.
Groups:
- Ziprasidone HCl (Zeldox): Ziprasidone hydrochloride (HCl) dosed according to the approved indications for disease diagnosis per local product document
Period: Overall Study
Arm/Group | Ziprasidone HCl (Zeldox)
Started | 3391
Completed | 3018
Not Completed | 373
Not completed — Adverse Event | 64
Not completed — Other | 309

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 3391
Age, Customized [Number; unit: participants]
  <18 years | 105
  Between 18 and 44 years | 2377
  Between 45 and 64 years | 723
  >=65 years | 186
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1926
  Male | 1465
Clinical Global Impression of Severity (CGI-S) status - Intent to treat population (ITT) [Number; unit: participants] — Single-item clinician rated scale to rate severity of illness over time. Scores range 1 (normal, not ill at all) to 7 (among the most extremely ill); higher score=more affected. ITT=administered at least 1 dose of study treatment at least once a week and observed for at least 1 efficacy assessment. N=participants with evaluable data at observation.
  participants
    Normal, not ill at all | 6
    Borderline mentally ill | 110
    Mildly ill | 669
    Moderately ill | 1264
    Markedly ill | 808
    Severely ill | 440
    Among the most extremely ill | 54
CGI-S status - Per protocol population (PP) [Number; unit: participants] — Single-item clinician rated scale to rate severity of illness over time. Scores range 1 (normal) to 7 (among the most extremely ill); higher score=more affected. PP= ITT group, study treatment for at least 8 (± 1 week) since enrollment, observed for final efficacy (inpatient visit, phone call). N=participants with evaluable data at observation.
  participants
    Normal, not ill at all | 3
    Borderline mentally ill | 68
    Mildly ill | 454
    Moderately ill | 877
    Markedly ill | 547
    Severely ill | 266
    Among the most extremely ill | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Clinical Global Impression of Severity (CGI-S) Status at Final Visit (up to Week 8) - Intent to Treat Population
Description: CGI-S is a single-item clinician rated scale to rate the severity of a participant's illness over time. Scores range from 1 (normal, not ill at all) to 7 (among the most extremely ill); higher score indicates more affected.
Time Frame: Baseline up to Week 8
Population: Intent to treat population (ITT): administered at least 1 dose of study treatment at least once a week and observed for at least 1 efficacy assessment. N=number of participants with evaluable data at observation. Efficacy analysis planned for CGI-S at each visit but completed at last visit (no set schedule for study visits).
Measure: Number; unit: particpants
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 3351
particpants
  Normal, not ill at all | 190
  Borderline mentally ill | 1125
  Mildly ill | 1325
  Moderately ill | 506
  Markedly ill | 156
  Severely ill | 46
  Among the most extremely ill | 3

2. Primary Outcome: Number of Participants for Clinical Global Impression of Severity (CGI-S) Status at Final Visit (up to Week 8) - Per Protocol Population
Description: as for outcome 1
Time Frame: Baseline up to Week 8
Population: Per Protocol population (PP): participants in ITT group with study treatment for at least 8 (± 1 week) since enrollment and observed for final efficacy (inpatient visit or phone call). N=participants with evaluable data at observation. Efficacy analysis planned for CGI-S at each visit but completed at last visit (no set schedule for study visits).
Measure: Number; unit: participants
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 2254
participants
  Normal, not ill at all | 130
  Borderline mentally ill | 815
  Mildly ill | 889
  Moderately ill | 320
  Markedly ill | 77
  Severely ill | 21
  Among the most extremely ill | 2

3. Primary Outcome: Number of Participants for Change From Baseline in Clinical Global Impression - Improvement (CGI-I) at Final Visit (up to Week 8) - ITT
Description: CGI-I is a single-item clinician rated scale used to assess the participant's improvement or worsening from baseline. Scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse); higher score indicates more affected.
Time Frame: Baseline up to Week 8
Population: ITT; N=number of participants with evaluable data at observation. Efficacy analysis planned for CGI-I at each visit but completed at last visit (no set schedule for study visits).
Measure: Number; unit: participants
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 3351
participants
  Very much improved | 368
  Much improved | 1026
  Minimally improved | 1361
  No change | 512
  Minimally worse | 71
  Much worse | 13
  Very much worse | 0

4. Primary Outcome: Number of Participants for Change From Baseline in Clinical Global Impression - Improvement (CGI-I) at Final Visit (up to Week 8) - PP
Description: as for outcome 3
Time Frame: Baseline up to Week 8
Population: PP; N=number of participants with evaluable data at observation. Efficacy analysis planned for CGI-I at each visit but completed at last visit (no set schedule for study visits).
Measure: Number; unit: participants
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 2254
participants
  Very much improved | 271
  Much improved | 751
  Minimally improved | 889
  No change | 299
  Minimally worse | 36
  Much worse | 8
  Very much worse | 0

5. Other Pre Specified Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS ) - Improvement
Description: BPRS-A: 18-item clinician rated scale to assess somatic concern, anxiety, emotional withdrawal, disorganization, hallucinatory behavior, guilt feelings, suspiciousness, disorientation, tension, mannerisms, posturing, grandiosity, depressive mood, hostility, motor retardation, uncooperativeness, unusual thought content, blunted affect, and excitement. Ratings anchored to improve consistency for a single rater over time or between raters. Items rated on 7-point scale 0 (not present) to 6 (extremely severe). Total score=sum of items (range 0 to 108); higher scores indicate increased pathology.
Time Frame: Baseline up to Week 8
Population: Safety analysis set: all participants who received at least 1 dose of study treatment. It was recommended to use the optional BPRS tool to gather additional information for the improvement score under usual practice. The optional BPRS tool was not used during the study.
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Change From Baseline in Drug Attitude Inventory (DAI-10) - Improvement
Description: DAI-10: a 10-item scale to assess how the attitude of participants with schizophrenia toward their medications may affect compliance. Respondents indicate 'true' or 'false' for each item. An overall calculated score ranges from -10 to 10, where a positive score indicates a positive subjective response (compliant); a negative score indicates non-compliance.
Time Frame: Baseline up to Week 8
Population: Safety analysis set. It was recommended to use the optional DAI-10 tool to gather additional information for the improvement score under usual practice. The optional DAI-10 tool was not used during the study.
Arm/Group | Ziprasidone HCl (Zeldox)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Ziprasidone HCl (Zeldox)
Serious Adverse Events (participants affected / at risk) | 2/3391
Other Adverse Events (participants affected / at risk) | 392/3391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone HCl (Zeldox) (N=3391)
Asthenia (General disorders) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone HCl (Zeldox) (N=3391)
Leukopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 24
Salivary hypersecretion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 33
Drug ineffective (General disorders) | 2
Gait disturbance (General disorders) | 3
Pyrexia (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Polydipsia (Metabolism and nutrition disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Akathisia (Nervous system disorders) | 80
Dizziness (Nervous system disorders) | 26
Dysarthria (Nervous system disorders) | 3
Dystonia (Nervous system disorders) | 14
Extrapyramidal disorder (Nervous system disorders) | 68
Headache (Nervous system disorders) | 20
Hypertonia (Nervous system disorders) | 2
Hypokinesia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 2
Motor dysfunction (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 72
Tremor (Nervous system disorders) | 12
Visual field defect (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 39
Blunted affect (Psychiatric disorders) | 1
Drug dependence (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 58
Schizophrenia (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 2
Thinking abnormal (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Nocturia (Psychiatric disorders) | 1
Mammary duct ectasia (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 2
Oculogyric crisis (Eye disorders) | 1
Vision blurred (Eye disorders) | 6

LIMITATIONS AND CAVEATS:
Per the Statistical Analysis Plan Amendment CGI-S and CGI-I endpoints analyzed as frequency counts (categorical) rather than the planned CGI-S mean change from baseline and CGI-I mean scores (continuous); any additional analyses would be exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.